CLINICAL TRIAL: NCT07384234
Title: SHR-1701 Combined With Chemotherapy for Gastric or Gastroesophageal Junction Adenocarcinoma With Peritoneal Metastasis: A Randomized, Two-Cohort Study
Brief Title: SHR-1701 Combined With Chemotherapy for Gastric or Gastroesophageal Junction Adenocarcinoma With Peritoneal Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-026
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Gastric Adenocarcinoma and Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — SHR-1701; Capecitabine; S 1 (combination); Paclitaxel; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1701 and intravenous/intraperitoneal paclitaxel and S-1 (Experimental)
  Interventions: Drug: SHR-1701; Drug: S-1; Drug: Paclitaxel
- SHR-1701 and CAPOX (Experimental)
  Interventions: Drug: SHR-1701; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: SHR-1701 — SHR-1701, 1800mg, Q3w
Drug: Capecitabine — Capecitabine, Q3W
  Arms: SHR-1701 and CAPOX
Drug: S-1 — S-1, Q3W
  Arms: SHR-1701 and intravenous/intraperitoneal paclitaxel and S-1
Drug: Paclitaxel — Paclitaxel,Q3W
  Arms: SHR-1701 and intravenous/intraperitoneal paclitaxel and S-1
Drug: Oxaliplatin — Oxaliplatin, Q3W
  Arms: SHR-1701 and CAPOX

SUMMARY:
This study is a prospective, randomized, two-cohort trial designed to evaluate the efficacy and safety of two regimens in the treatment of gastric or gastroesophageal junction adenocarcinoma with peritoneal metastasis: SHR-1701 combined with intravenous and intraperitoneal paclitaxel plus S-1, or SHR-1701 combined with CAPOX.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Pathologically confirmed gastric or gastroesophageal junction adenocarcinoma (Siewert typeⅡ and type Ⅲ gastroesophageal junction adenocarcinoma are eligible for inclusion).
3. Definitively diagnosed with peritoneal metastasis by exploratory laparoscopy and/peritoneal lavage cytology (CY0P1/CY1P0/CY1P1 are eligible, ovarian metastasis is permitted), and without gastric outlet obstruction or intestinal obstruction.
4. No prior anti-tumor treatment history (including radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.).
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
6. Normal function of major organs.

Exclusion Criteria:

1. Known HER2-positive.
2. Previous history of gastric cancer surgery.
3. Contraindications to surgical treatment or chemotherapy, or poor physical status and organ function precluding major abdominal surgery.
4. Presence of distant metastases other than peritoneal metastases (e.g., liver, lung, ovarian, para-aortic lymph node, brain metastases, etc.).
5. Active autoimmune disease within 4 weeks prior to enrollment or a history of autoimmune disease.
6. Significant cardiovascular disease within 6 months prior to enrollment, including unstable angina or myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival rate | Up to 2 years

SECONDARY OUTCOMES:
Conversion surgery rate | Up to 4 weeks after completion of surgery
R0 resection rate | Up to 4 weeks after completion of surgery
Pathological complete response(pCR) | Up to 4 weeks after completion of surgery
Tumor regression grade | Up to 4 weeks after completion of surgery
Event free survival (EFS) | Up to 2 years
DFS | Up to 2 years
  Disease-free survival (DFS)
Overall survival(OS) | Up to 3 years
AEs | Up to approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanan Zheng, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No